CLINICAL TRIAL: NCT06858657
Title: A Single and Multiple Ascending Dose Study to Assess the Safety,Tolerability, PK,PD and Food Effect of HSK44459 in Healthy Subjects
Brief Title: A Phase I Study to Assess the Safety,Tolerability, PK, PD, and Food Effect of HSK44459 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Haisco Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSK44459-101
Record Dates: First submitted 2024-08-15; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: HSK44459; healthy subjects; phase1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HSK4449 (Experimental): Single or multiple oral doses of HSK44459, and food effect of HSK44459
  Interventions: Drug: HSK44459
- Placebo (Placebo Comparator): Single or multiple oral doses of placebo, and food effect of placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: HSK44459 — Dose 1 to Dose 5
  Arms: HSK4449
Drug: placebo — dose 1 to dose 5
  Arms: Placebo

SUMMARY:
This is a Phase I, randomized, subject-blinded, placebo controlled study to assess the safety, tolerability, pharmacokinetic (PK), pharmacodynamic (PD),and food effect (FE) of HSK44459 following (1) a single ascending dose (part 1), (2) 10 days of multiple ascending dose (part 2), and (3) a single dose two-period crossover FE cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form, understand the trialprocedures, and be willing to comply with all trial procedures andrestrictions;
2. 18 years to 55 years (inclusive), male and female;
3. Male subjects weight ≥50 kg and female subjects weight ≥45 kg. Bodymass index (BMI) : 19-26 kg/m2 (inclusive) ;
4. Subjects are willing to voluntarily use effectivecontraceptives from screening to at least 3 months after the last dose administration.

Exclusion Criteria:

1. Have a history of severe and uncontrolled diseases, such ascardiovascular, respiratory, liver, gastrointestinal, endocrine,hematologic, mental/nervous systems diseases within 3 months prior to screening;
2. Have an infection that requires systematic treatment with antibiotics, antifungal, antiparasitic or antiviral drugs;
3. Have a history of any malignant tumors;
4. The abnormalities were clinically significant during the screening period, such as physical examination, vital signs, blood biochemistry, blood routine, coagulation, urine routine, blood pregnancy test, infectious diseases and X-ray;
5. Subjects whose results of routine 12-lead electrocardiograms were inconsistent with normal heart conduction and function;
6. Previous or current gastrointestinal, liver, kidney, or other disease known to interfere with drug absorption, distribution, metabolism, or excretion;
7. Smoking more than 5 cigarettes per day within 3 months prior toscreening or smoking during the study;
8. Average alcohol intake is more than 14 unit per week (1unit=10g alcohol , 1 unit=285 mL 4.9% alcohol beer, or 30 mL 40% alcohol spirit, or 100mL 12% alcohol wine) within the 3 months prior to screening, or positive urine drug screen at screening;
9. Have a history of high consumption of grapefruit juice, methylxanthinerich food or beverage (such as coffee, tea, cola, chocolate, energydrinks) ,consumption of grapefruit juice;
10. Blood donation (or blood loss) ≥400 mL, or receiving blood products to improve anemia within 3 months prior to the screening;
11. Subjects who have a allergic to any component of HSK44459 or allergic history to opiates;
12. Have participated in any clinical investigator within 3 months prior to screening;
13. A pregnant/lactating woman, or has a positive pregnancy test at screening or during the trial;
14. Not suitable for this study as judged by the investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2024-08-17 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-20 (Actual)

PRIMARY OUTCOMES:
The number and severity of treatment emergent adverse events (TEAEs) | 7 days after single dose and 3 days after the first dose of multiple doses
  To assess the safety and tolerability of single or multiple oral dose of HSK44459 in healthy adult volunteers

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, China

IPD SHARING:
Plan to Share IPD: No